CLINICAL TRIAL: NCT05997823
Title: Is Dorso-Volar Kinesiotape Added to the Home Exercise Program Effective in the Treatment of Carpal Tunnel Syndrome?-Prospective Randomized Controlled Study
Brief Title: Dorsovolar Kinesiotape in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Asst. Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/11-08
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome Treatment
Keywords: carpal tunnel syndromes; kinesiotape; electromyography; median neuropathy; muscle strength; pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Pain | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- home exercises (Active Comparator)
  Interventions: Other: home exercises
- sham-KT and home exercises (Experimental)
  Interventions: Other: kinesiotape; Other: home exercises
- dorso-volar KT and home exercises (Experimental)
  Interventions: Other: kinesiotape; Other: home exercises

INTERVENTIONS:
Other: kinesiotape — The button hole technique was used for area correction during the KT application (Figure 1). Two I-tapes were applied, one from the medial epicondyle to the proximal phalanx on the palmar side and the other from the lateral epicondyle to the proximal phalanx on the dorsal side. The area where the phalanges are located was marked, and two hole was drilled in the center.After cleaning the skin with alcohol, the tape to be applied to the palmar side was passed over the 3rd and 4th fingers, and the patient was asked to perform radial deviation and wrist extension
  Arms: dorso-volar KT and home exercises; sham-KT and home exercises
Other: home exercises — home exercises

SUMMARY:
This study aimed to compare the short- and medium-term efficacy of dorso-volar kinesiotape (KT) added to home exercises (HE) with sham-KT and HE alone in the treatment of mild or moderate carpal tunnel syndrome (CTS) in terms of pain, symptom severity, function, grip strength, and electrophysiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* pain or numbness radiating to the palm for at least 6 weeks,
* at least one positive Tinel's, Phalen's, or carpal compression test on physical examination, and
* mild/moderate CTS on EMG examination.

Exclusion Criteria:

* Metabolic disease (diabetes, rheumatoid arthritis, thyroid disease),
* systemic or malignant disease, history of trauma, fracture or surgery to the wrist,
* physical therapy programs, surgical procedures, injections or KT applications to the wrist for CTS treatment in the past year,
* severe thenar atrophy,
* C6-C7 radiculopathy among CTS differential diagnoses,
* cervical spondylosis, thoracic outlet syndrome, entrapment of the median nerve above the wrist,
* polyneuropathy or traumatic injury to the median nerve,
* rashes or open wounds on the skin of the wrist and forearm that could prevent treatment with kinesiology taping

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Electrodiagnostic Evaluation | 30 minutes
  Superficial recording electrodes were placed in the abductor pollicis brevis (APB) muscles (recording stimulus distance 5 cm) for median nerve motor conduction and in the abductor digiti minimi (ADM) muscles (recording stimulus distance 5 cm) for ulnar nerve motor conduction.Superficial recording electrodes were placed on the 3rd finger for median nerve sensory conduction (recording stimulus distance 13 cm) and on the 5th finger for ulnar nerve sensory conduction (recording stimulus distance 11 cm).The ground electrode was placed between the recording and stimulus electrodes for all electrophysiological tests.Sensory latency, amplitude, and conduction velocity of the median nerve and motor latency, amplitude, and conduction velocity were recorded
Hand Strength | 10 minutes
  A Jamar hand dynamometer (Baseline ® hydraulic hand dynamometer, Irvington, NY, USA) was used to measure handgrip strength.
Pain Evaluation | 5 minutes
  A 10-point visual analog scale (VAS) was used to rate pain. Patients were asked to rate the pain they felt at rest, at night, and with movement with a number ranging from 0 (no pain) to 10 (very severe), VAS movement, VAS night, and VAS rest
Finger Strength | 10 minutes
  A pinch meter (Baseline ® hydraulic pinch gauge, Irvington, NY, USA) was used to evaluate lateral grip strength (LGS) and pinch grip strength

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Kocaeli Derince Training and Research Hospital, Kocaeli, Deince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No